CLINICAL TRIAL: NCT04570410
Title: Trials of Primary Excision Combined With Preoperative Neoadjuvant Therapy and Adjuvant Therapy Was Used as a First-line Comprehensive Therapy for Oligometastasis of Urothelial Carcinoma（UC）.
Brief Title: Primary Excision Combined With Preoperative Neoadjuvant and Adjuvant Therapy for Oligometastasis of Urothelial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-SR-264.A1
Record Dates: First submitted 2020-09-16; First posted 2020-09-30 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-04

CONDITIONS: Bladder Urothelial Carcinoma
Keywords: Oligometastasis; PD-1; Gemcitabine plus cisplatin; Simple lymph node metastasis
MeSH Terms: interventions — Lymph Node Excision; tislelizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GC plus Tislelizumab combined with RC (Experimental): GC plus Tislelizumab Participants receive GC (Gemcitabine plus cisplatin), in combination with Tislelizumab administered intravenously (IV) every 3 weeks (Q3W) before surgery.Immunotherapy was continued for 12 months after excision of the primary lesion.
  Intervention/treatment： Biological: Tislelizumab Tislelizumab IV infusion of 200 mg Q3W
  Biological: GC GC (Gemcitabine plus cisplatin): Gemcitabine 1000mg/m2 D1,D8 iv every 3 weeks Cisplatin70mg/m2,D2,3,4 iv every 3 weeks
  Interventions: Procedure: primary focal resection plus lymph node dissection; Drug: Tislelizumab; Drug: Gemcitabine plus cisplatin

INTERVENTIONS:
Procedure: primary focal resection plus lymph node dissection — Primary radical resection plus lymph node dissection was performed in patients with oligometastatic urothelial carcinoma
Drug: Tislelizumab — Tislelizumab IV infusion of 200 mg Q3W
  Other Names: PD-1
Drug: Gemcitabine plus cisplatin — GC (Gemcitabine plus cisplatin): Gemcitabine 1000mg/m2 D1,D8 iv every 3 weeks Cisplatin70mg/m2,D2,3,4 iv every 3 weeks
  Other Names: GC

SUMMARY:
treatment of primary focal resection plus lymph node dissection combined with chemotherapy and anti-programmed cell death 1(PD-1) for Oligometastasis of urothelial carcinoma.

DETAILED DESCRIPTION:
The study is designed to demonstrate that Whether the perioperative comprehensive treatment of primary focal resection plus lymph node dissection combined with chemotherapy and anti-PD-1 can prolong the overall survival of patients, narrow the range of metastatic lesions and improve the quality of life of patients.

Compared with patients with extensive metastasis, 2-year tumor-specific survival and overall survival of patients with oligometastatic bladder cancer were significantly increased (53.3% vs 16.1%)；(51.9% vs. 15.4%).Gemcitabine plus cisplatin (GC) regimen has been shown to bring clinical benefits in neoadjuvant therapy of metastatic UC（urothelial carcinoma）.

PD-1 inhibitors have been widely used in urothelial carcinoma in recent years, and positive data have been obtained in both advanced patients and neoadjuvant patients.

If successful in this trial, it will serve to provide a therapeutic alternative for this patient who have oligometastasis of urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oligometastatic urothelial carcinoma, including :patients with T2-T4 with any metastasis urothelial carcinoma diagnosed by pathology and evaluated by imaging. 1. Patients with measurable oligometastasis or with local lymph node metastasis. Measurable oligometastasis includes: A. a solitary metastatic organ, B. number of metastatic lesions of ≤3, C. the largest diameter of metastatic foci of ≤5cm, D. absence of liver metastasis. 2. Local lymph node metastasis includes: M0 patients with the short diameter of pelvic lymph nodes was ≥8 mm. The researchers assessed the benefits of excision of the primary lesion.
* Older than 18 years old.
* Volunteer to participate in the trial, be able to provide a written informed consent, and understand and agree to comply with the study requirements and evaluation schedule.
* Eastern Cooperative Oncology Group (ECOG) performance status <2
* International standardized ratio or activated partial thrombin time ≤1.5 upper limit of normal value (ULN);The calculated creatinine clearance rate was ≥60ml/min;Serum total bilirubin ≤1.5×ULN;aspartate transaminase(AST), Alanine transaminase(ALT) and alkaline phosphatase ≤2.5×ULN;
* Non-pregnant or fertile men or women must be willing to take effective contraceptive measures during the study period and ≥120 days after the last administration of tislelizumab, and the women should be negative on urine or serum pregnancy test results less than or equal to 7 days before enrollment.

Exclusion Criteria:

* Previous therapy targeted at PD-1, PD-L1, PD-L2, Cytotoxic T-Lymphocyte Associated Protein 4(CTLA-4)or other antibodies or drugs specifically targeting T cell synergistic stimulation or checkpoint channels.
* Other approved systemic anti-cancer therapies or systemic immune modulators (including but not limited to interferon, interleukin-2, and tumor necrosis factor) were received within 28 days prior to enrollment.
* Severe chronic or active infections requiring systemic antimicrobial, antifungal, or antiviral therapy within 14 days prior to enrollment.
* Major surgery or major trauma occurred within 28 days prior to enrollment.
* Live vaccine was administered within 28 days before enrollment.
* Received any herbal or proprietary Chinese medicine used to control cancer in the 14 days prior to enrollment.
* Active autoimmune disease requiring long-term use of large amounts of hormones and other immunosuppressive agents.
* The researchers identified abnormalities in potassium, sodium, calcium, or hypoalbuminemia, interstitial lung disease, non-infectious pneumonia, or other uncontrolled whole-body diseases, including diabetes, hypertension, and cardiovascular disease, that may affect treatment.
* A history of HIV, hepatitis B virus(HBV)and hepatitis C virus(HCV) infection is known.
* A history of known allergic reactions to any of the drugs studied.
* Is participating in additional clinical studies.
* The researcher believes that the patient is not suitable to participate in this study (such as the treatment that does not meet the patient's greatest benefit, patient compliance, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Pathological complete response (ypT0N0) | From treatment to surgery
  Pathological confirmation is ypT0N0

SECONDARY OUTCOMES:
Pathological downstaging | From treatment to surgery
  Pathological confirmation is <ypT2N0
progression-free survival(PFS) | through study completion, an average of 1 year
  time between the first objective recording of PD(progressive disease) or death from any cause (whichever occurs first) from first treatment.
Overall survival (OS) | through study completion, an average of 1 year
  time between death (any causes) from first treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Lv, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The first affiliated hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erratum: Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2020 Jul;70(4):313. doi: 10.3322/caac.21609. Epub 2020 Apr 6. No abstract available. PMID 32767693
- [Background] Rosenberg JE, Carroll PR, Small EJ. Update on chemotherapy for advanced bladder cancer. J Urol. 2005 Jul;174(1):14-20. doi: 10.1097/01.ju.0000162039.38023.5f. PMID 15947569
- [Background] Bajorin DF, Dodd PM, Mazumdar M, Fazzari M, McCaffrey JA, Scher HI, Herr H, Higgins G, Boyle MG. Long-term survival in metastatic transitional-cell carcinoma and prognostic factors predicting outcome of therapy. J Clin Oncol. 1999 Oct;17(10):3173-81. doi: 10.1200/JCO.1999.17.10.3173. PMID 10506615
- [Background] Hellman S, Weichselbaum RR. Oligometastases. J Clin Oncol. 1995 Jan;13(1):8-10. doi: 10.1200/JCO.1995.13.1.8. No abstract available. PMID 7799047
- [Background] Seisen T, Sun M, Leow JJ, Preston MA, Cole AP, Gelpi-Hammerschmidt F, Hanna N, Meyer CP, Kibel AS, Lipsitz SR, Nguyen PL, Bellmunt J, Choueiri TK, Trinh QD. Efficacy of High-Intensity Local Treatment for Metastatic Urothelial Carcinoma of the Bladder: A Propensity Score-Weighted Analysis From the National Cancer Data Base. J Clin Oncol. 2016 Oct 10;34(29):3529-3536. doi: 10.1200/JCO.2016.66.7352. PMID 27269944
- [Background] Dong F, Shen Y, Gao F, Xu T, Wang X, Zhang X, Zhong S, Zhang M, Chen S, Shen Z. Prognostic value of site-specific metastases and therapeutic roles of surgery for patients with metastatic bladder cancer: a population-based study. Cancer Manag Res. 2017 Nov 14;9:611-626. doi: 10.2147/CMAR.S148856. eCollection 2017. PMID 29180897
- [Background] Horwich A, Babjuk M, Bellmunt J, Bruins HM, De Reijke TM, De Santis M, Gillessen S, James N, Maclennan S, Palou J, Powles T, Ribal MJ, Shariat SF, Van Der Kwast T, Xylinas E, Agarwal N, Arends T, Bamias A, Birtle A, Black PC, Bochner BH, Bolla M, Boormans JL, Bossi A, Briganti A, Brummelhuis I, Burger M, Castellano D, Cathomas R, Chiti A, Choudhury A, Comperat E, Crabb S, Culine S, De Bari B, DeBlok W, De Visschere PJL, Decaestecker K, Dimitropoulos K, Dominguez-Escrig JL, Fanti S, Fonteyne V, Frydenberg M, Futterer JJ, Gakis G, Geavlete B, Gontero P, Grubmuller B, Hafeez S, Hansel DE, Hartmann A, Hayne D, Henry AM, Hernandez V, Herr H, Herrmann K, Hoskin P, Huguet J, Jereczek-Fossa BA, Jones R, Kamat AM, Khoo V, Kiltie AE, Krege S, Ladoire S, Lara PC, Leliveld A, Linares-Espinos E, Logager V, Lorch A, Loriot Y, Meijer R, Carmen Mir M, Moschini M, Mostafid H, Muller AC, Muller CR, N'Dow J, Necchi A, Neuzillet Y, Oddens JR, Oldenburg J, Osanto S, Oyen WJG, Pacheco-Figueiredo L, Pappot H, Patel MI, Pieters BR, Plass K, Remzi M, Retz M, Richenberg J, Rink M, Roghmann F, Rosenberg JE, Roupret M, Rouviere O, Salembier C, Salminen A, Sargos P, Sengupta S, Sherif A, Smeenk RJ, Smits A, Stenzl A, Thalmann GN, Tombal B, Turkbey B, Vahr Lauridsen S, Valdagni R, Van Der Heijden AG, Van Poppel H, Vartolomei MD, Veskimae E, Vilaseca A, Vives Rivera FA, Wiegel T, Wiklund P, Williams A, Zigeuner R, Witjes JA. EAU-ESMO consensus statements on the management of advanced and variant bladder cancer-an international collaborative multi-stakeholder effort: under the auspices of the EAU and ESMO Guidelines Committeesdagger. Ann Oncol. 2019 Nov 1;30(11):1697-1727. doi: 10.1093/annonc/mdz296. PMID 31740927
- [Background] Ogihara K, Kikuchi E, Watanabe K, Kufukihara R, Yanai Y, Takamatsu K, Matsumoto K, Hara S, Oyama M, Monma T, Masuda T, Hasegawa S, Oya M. Can urologists introduce the concept of "oligometastasis" for metastatic bladder cancer after total cystectomy? Oncotarget. 2017 Dec 4;8(67):111819-111835. doi: 10.18632/oncotarget.22911. eCollection 2017 Dec 19. PMID 29340094